CLINICAL TRIAL: NCT00257764
Title: A Randomised Controlled Trial of Dysphagia Therapies for Swallowing Disorders Following Stroke.
Brief Title: Behavioural Intervention for Dysphagia in Acute Stroke
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Royal Perth Hospital (Other)
Collaborators: Royal Perth Hospital Medical Research Foundation (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RPH00096
Record Dates: First submitted 2005-11-21; First posted 2005-11-23 (Estimated); Last update posted 2006-05-05 (Estimated); Status verified 1999-06

CONDITIONS: Dysphagia
Keywords: Swallowing disorder; Stroke; Standardized swallowing therapy; Randomized controlled trial
MeSH Terms: conditions — Deglutition Disorders; Stroke

INTERVENTIONS:
Behavioral: behavioral swallowing exercises/ strategies

SUMMARY:
Swallowing dysfunction after stroke is common, but there is no reliable evidence for how it should be managed other than perhaps by nasogastric tube. This study compared the effectiveness of standardised, low and high intensity behavioral intervention for dysphagia with that of "usual care".

DETAILED DESCRIPTION:
Stroke compromises swallowing function, causing dysphagia, in one quarter to one half of all patients. Dysphagia is associated with an increased risk of aspiration pneumonia, dehydration and malnutrition. Despite the development and implementation of several strategies of managing dysphagia after stroke, Few have been evaluated by means of randomised controlled trials.

Comparisons: This study aims to compare stroke patients with dysphagia assigned to receive usual swallowing care, prescribed by the attending physician; standardised low intensity intervention comprising swallowing compensation strategies and diet prescription; or standardised high intensity intervention and dietary prescription .

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of stroke within the previous 7 days
* clinical diagnosis of swallowing difficulty

Exclusion Criteria:

* no previous history of swallowing treatment
* no previous history of surgery of the head or neck

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 1996-05; Study Completion 1999-05

PRIMARY OUTCOMES:
survival free of an abnormal diet at 6 months

SECONDARY OUTCOMES:
time to return to normal diet over the study
recovery of swallowing ability at 6 months after stroke
the occurrence of dysphagia - related medical complications at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Graeme Hankey, MBBS, MD,, Study Director — Royal Perth Hospital; Giselle D Mann, MPH,PhD, Principal Investigator — Royal Perth Hospital
Locations (1):
- Royal Perth Hospital, Perth, Western Australia, Australia

REFERENCES:
- [Result] Carnaby G, Hankey GJ, Pizzi J. Behavioural intervention for dysphagia in acute stroke: a randomised controlled trial. Lancet Neurol. 2006 Jan;5(1):31-7. doi: 10.1016/S1474-4422(05)70252-0. PMID 16361020